CLINICAL TRIAL: NCT01000220
Title: Evaluation of Omeprazole Effect on Glaucoma
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shahid Beheshti University of Medical Sciences (Other)
Collaborators: Ophthalmic Research Center (Ambiguous)
Responsible Party: Ophthalmic Research Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 8735
Record Dates: First submitted 2009-07-07; First posted 2009-10-22 (Estimated); Last update posted 2010-05-04 (Estimated); Status verified 2009-10

CONDITIONS: Glaucoma
MeSH Terms: conditions — Glaucoma | interventions — Omeprazole

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Omeprazole (Active Comparator)
  Interventions: Drug: Omeprazole
- placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Omeprazole
  Arms: Omeprazole
Drug: Placebo
  Arms: placebo

SUMMARY:
Omeprazole is a safe drug listed in OTC drug due to its safety. It acts by irreversible inhibition of K/H ATP ase pump and also Na/K ATP ase, Na/H ATP ase.Considering these actions the effect of omeprazole on decreasing intra ocular pressure is an issue of debate.In this Randomized Clinical Trial conducted in labafinejad hospital, patients with glaucoma who need to take omeprazole due to GI problem are evaluated in two groups including placebo and drug users. The effect will be finally assessed.

DETAILED DESCRIPTION:
Omeprazole is a safe drug listed in OTC drug due to its safety. It acts by irreversible inhibition of K/H ATP ase pump and also Na/K ATP ase, Na/H ATP ase.Considering these actions the effect of omeprazole on decreasing intra ocular pressure is an issue of debate.In this Randomized Clinical Trial conducted in labafinejad hospital, patients with glaucoma who need to take omeprazole due to GI problem are evaluated in two groups including placebo and drug users. The effect will be finally assessed.

ELIGIBILITY:
Inclusion Criteria:

* patients with glaucoma
* 18 to 70 years
* POAG patients, Pseudoexfoliation
* no history of other systemic disease
* no history of intraocular intervention
* no history of H2 blocker or PPI consumption during the past month consuming 2 or less topical anti-glaucoma medication
* no present immune deficiency
* no addiction habit

Exclusion Criteria:

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Locations (1):
- Ophthalmic Research Center, Tehran, Tehran Province, Iran